CLINICAL TRIAL: NCT07274059
Title: Clinical Study on the Safety and Efficacy of Allogeneic, Umbilical Cord Blood Derived CAR T-cell Therapy for Refractory Systemic Lupus Erythematosus
Brief Title: Allogeneic UCB-derived CAR-T for SLE
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chengdu Ucello Biotechnology Co., Ltd. (Industry)
Collaborators: The General Hospital of Western Theater Command (Other); Yancheng Third People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UDCAR-SLE
Record Dates: First submitted 2025-11-22; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: SLE - Systemic Lupus Erythematosus
Keywords: allogeneic; CAR-T; umbilical cord blood; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — bis(3-bis(4-chlorophenyl)methyl-4-dimethylaminophenyl)amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UCAR-T cells treatment (Experimental)
  Interventions: Drug: allogeneic umbilical cord blood-derived CAR-T targeting CD19 and BCMA

INTERVENTIONS:
Drug: allogeneic umbilical cord blood-derived CAR-T targeting CD19 and BCMA — intravenous injection of allogeneic umbilical cord blood-derived CAR-T targeting CD19 and BCMA

SUMMARY:
The purpose of this clinical trial is to learn if allogeneic, umbilical cord blood-derived chimeric antigen receptor T-cell (UCAR-T) targeting CD19 and BCMA works to treat refractory SLE in adults. It will also learn about the safety and efficacy of the UCAR-T cell product.

DETAILED DESCRIPTION:
* The main questions it aims to answer are: What CAR-T-related adverse events (AEs) occur within 3 months after the UCAR-T cell infusion? Which dose level is the optimal biological dose (OBD)? What are the changes of disease activity status, proportion of patients achieving DORIS remission, percentage of participants achieving maintenance of drug-free DORIS remission, proportion of patients achieving SRI-4 remission, percentage of participants achieving maintenance of LLDAS?
* Participants will may receive lymphodepletion chemotherapy (fludarabine plus cyclophosphamide) if clinically needed. If lymphodepletion chemotherapy is administered, rest for 2 days on Day -2 and Day -1. Receive UCAR-T cells infusion on Day 0. Then be hospitalized for at least 7 days post-infusion for close safety monitoring and remain within 2 hours of the treatment facility for at least 28 days. Visit the clinic at Day 14, Day 28, month 3, month 6, month 9, month 12, month 18 and month 24 after UCAR-T cells infusion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years (inclusive), regardless of gender.
* Definitive diagnosis of systemic lupus erythematosus (SLE) meeting the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria for SLE
* Treatment refractory: failed ≥ 2 conventional SLE treatments for at least 3 months.
* Disease activity assessed by SELENA-SLEDAI score ≥ 6 with at least one British Isles Lupus Assessment Group (BILAG)-2004 Class A (severe manifestation) or two Class B (moderate manifestation) organ scores (or both); OR SELENA-SLEDAI score ≥ 8.
* Adequate function of major organs as follows:

Bone marrow function: a. Neutrophil count ≥ 1 × 10⁹/L (no colony-stimulating factor therapy within 2 weeks prior to testing, excluding neutropenia caused by SLE); b. Hemoglobin ≥ 60 g/L.

Liver function: Alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN) (excluding ALT elevation caused by SLE); Aspartate aminotransferase (AST) ≤ 3 × ULN (excluding AST elevation caused by SLE); Total bilirubin (TBIL) ≤ 1.5 × ULN (excluding TBIL elevation caused by SLE).

Renal function: Creatinine clearance rate (CrCl) ≥ 30 mL/minute (calculated by Cockcroft/Gault formula, excluding CrCl reduction caused by SLE).

Coagulation function: International normalized ratio (INR) ≤ 1.5 × ULN; Prothrombin time (PT) ≤ 1.5 × ULN.

Cardiac function: Hemodynamically stable.

* Female subjects of childbearing potential and male subjects whose partners are of childbearing potential must use medically approved contraceptive methods or abstain from sexual intercourse during the study treatment period and for at least 6 months after the end of study treatment. Female subjects of childbearing potential must have a negative serum human chorionic gonadotropin (HCG) test within 7 days prior to study enrollment and must not be breastfeeding.
* Voluntarily agrees to participate in the clinical study, signs the informed consent form (ICF), and demonstrates good compliance with study procedures and follow-up.

Exclusion Criteria:

* History of severe drug allergies or atopic diathesis.
* Presence or suspicion of uncontrolled or treatment-requiring fungal, bacterial, viral, or other infections.
* Cardiac function insufficient to tolerate the study treatment.
* Congenital immunoglobulin deficiency.
* History of malignant tumors within the past 5 years.
* End-stage renal failure.
* Positive for hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA titer above the lower limit of detection; positive for hepatitis C virus (HCV) antibody with positive peripheral blood HCV RNA; positive for human immunodeficiency virus (HIV) antibody; positive syphilis test.
* History of mental illness or severe cognitive impairment.
* Use of disease-modifying immunosuppressive agents within 5 half-lives or biological agents within 4 weeks prior to enrollment.
* Pregnant females or females planning to become pregnant.
* Other conditions deemed by the investigator to preclude study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence rate of Dose limited toxicity (DLTs) | Up to 28 days after infusion
  Dose limited toxicity(DLT) was defined as the occurrence of any of the following adverse events within 28 days of the infusion of UCAR-T cells.
the rate of adverse events | up to 2 months after UCAR-T injection
  The number, frequency, severity, and laboratory findings of all treatment-related adverse events/serious adverse events are included.

SECONDARY OUTCOMES:
Proportion of patients achieving DORIS remission | up to 2 years after UCAR-T injection
the changes of SELENA-SLEDAI score | up to 2 years after UCAR-T injection
Proportion of patients achieving SRI-4 remission | up to 2 years after UCAR-T injection
Percentage of participants achieving maintenance of drug-free DORIS remission | up to 2 years after UCAR-T injection
Percentage of participants achieving maintenance of LLDAS | up to 2 years after UCAR-T injection
the changes of BILANG 2004 score | up to 2 years after UCAR-T injection
  The BILAG 2004 score is a validated clinical assessment tool for systemic lupus erythematosus (SLE), which evaluates disease activity across 9 organ systems (constitutional, cutaneous, mucous membrane, musculoskeletal, renal, neurological, cardiovascular, respiratory, and hematological) using a 5-point grading scale (A=active/severe, B=active/mild-moderate, C=stable/minor activity, D=inactive, E=not involved) to guide treatment decisions and monitor therapeutic responses in clinical practice and research.
the changes of Physician's Global Assessment (PGA) | up to 2 years after UCAR-T injection

OTHER OUTCOMES:
AUC of CAR-T cells | up to 2 months after UCAR-T injection
  AUC is defined as the area under the curve in 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Wang, M.D., Principal Investigator — The General Hospital of Western Theater Command; Mei Dong Jiang, M.D., Principal Investigator — Yancheng Third People's Hospital
Locations (2):
- China (2):
  - Yancheng Third People's Hospital, Yancheng, Jiangsu
  - The General Hospital of Western Theater Command, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
The safety and efficacy data will be shared in a publication.
Time Frame: starting 6 months after publication